CLINICAL TRIAL: NCT00220168
Title: A Phase II Trial Evaluating Irinotecan and Capecitabine in Patients With Relapsed/Refractory Upper Gastrointestinal Tumours
Brief Title: Phase II Trial Evaluating Irinotecan and Capecitabine Relapsed/Refractory Upper GI Tumours
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Jane Lawrence, Royal Marsden NHS Foundation Trust
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2166
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Upper Gastrointestinal Tumours
MeSH Terms: interventions — Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Irinotecan, Capecitabine

SUMMARY:
The objective of this study is to assess the efficacy and toxicity of a 3 weekly regimen containing irinotecan combined with capecitabine in the setting of relapsed or refractory upper gastrointestinal tumours. Patients with locally advanced or metastatic adenocarcinoma or squamous cell carcinoma originating from the oesophagus, oesophagogastric junction or stomach who have previously received chemotherapy and have either failed to respond or who have relapsed within 3 months after an initial response will be eligible for treatment in this study.

The response rate, failure-free survival and overall survival of treated patients will be evaluated. Toxicity and quality of life will also be monitored closely.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma or squamous cell carcinoma of oesophagus, O-G junction and stomach, not amenable to surgical resection.
* Bidimensionally measurable disease, or unidimensional measurable disease assessable by CT scanning, not within previously irradiated areas.
* Patients with progressive disease during previous chemotherapy treatment or within three months of stopping treatment.
* At least one previous chemotherapy regimen, given within 3 months prior to inclusion in this study.
* No previous exposure to irinotecan.
* Adequate bone marrow function with platelets >100 X 109/L; WBC > 3 X 109/L; Neutrophils > 1.5 X 109/L at the time of study entry.
* Satisfactory renal function. Creatinine clearance (measured by Cockcroft and Gault) >50ml/min and Cr <135.
* Satisfactory liver function:
* In the absence of liver metastases: Bilirubin < 1.25N (N=upper limit of normal range) Hepatic transaminases < 2.5N Prothrombin time < 1.5N
* In the presence of liver metastases: Bilirubin < 1.5N Hepatic transaminases < 5N Prothrombin time < 1.5N
* No uncontrolled medical condition
* No previous malignant disease except for non-melanotic skin cancer or in-situ carcinoma of the uterine cervix.
* ECOG performance status of 0, 1 or 2.
* Predicted life expectancy of > 3 months.
* Adequate contraceptive precautions
* Informed written consent

Exclusion Criteria:

* Medical or psychiatric conditions resulting in inability of patient to give written consent.
* ECOG Performance status >2
* Intracerebral metastases or meningeal carcinomatosis
* Unresolved bowel obstruction
* Creatinine clearance <50ml/min, Cr >135
* Uncontrolled angina pectoris, heart failure (New York heart classification 3 or 4).
* Pregnancy/lactation
* Previous malignancy other than adequately treated basal cell carcinoma of the skin or cervical carcinoma in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2003-01

PRIMARY OUTCOMES:
Response rates
Time to disease progression (TTP)

SECONDARY OUTCOMES:
Survival
Quality of life
Toxicity (incidence of febrile neutropenia, in-patient admissions, severity of diarrhea, mucositis, aesthesia, transfusion requirements).

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom